CLINICAL TRIAL: NCT03455088
Title: The Effect of Dialectical Behavioral Group Therapy on the Patients With Bulimia Nervosa : A Multicenter Randomized Controlled Study
Brief Title: The Effect of G-DBT on the Patients With BN : A Multicenter Randomized Controlled Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Mental Health Center (Other)
Collaborators: Peking University Sixth Hospital (Other); Shanghai Tongji Hospital, Tongji University School of Medicine (Other)
Responsible Party: Principal Investigator, Jue CHEN, Director of Psychosomatic Department in Shanghai Mental Health Center, Shanghai Mental Health Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CRC2017YB02
Record Dates: First submitted 2018-02-11; First posted 2018-03-06 (Actual); Last update posted 2022-10-04 (Actual); Status verified 2022-10

CONDITIONS: Feeding and Eating Disorders
MeSH Terms: conditions — Feeding and Eating Disorders | interventions — Fluoxetine

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- DBT group (Experimental): DBT group has 55 patients, maybe will be divided them into 6 groups. Every group has 8-10 patients. Every group receive 12 times DBT group therapy and 1 times a week for 120 minutes each time.
  Interventions: Behavioral: Dialectical Behavioral Group Therapy
- Drug therapy group (Active Comparator): Drug therapy group has 55 patients, and the investigator may use fluoxetine as treatment drug.
  Interventions: Drug: Drug: fluoxetine
- DBT and drug therapy group (Experimental): DBT and drug therapy group has 55 patients, maybe the investigator can divide them into 7 groups. Every group has 8-10 patients. Every group receive 12 times DBT group therapy and 1 times a week for 120 minutes each time. At the same time, the investigator use fluoxetine as treatment drug.
  Interventions: Behavioral: Dialectical Behavioral Group Therapy; Drug: Drug: fluoxetine

INTERVENTIONS:
Behavioral: Dialectical Behavioral Group Therapy — DBT is based on the model for the development of emotion regulation, designed for teaching how to regulate their adaptive emotions and behaviors cased by mood disorders , so it is valid for BN patient.
  Arms: DBT and drug therapy group; DBT group
Drug: Drug: fluoxetine — Antidepressant fluoxetine can reduce binge eating and purging behaviors in BN patients in a short time.
  Arms: DBT and drug therapy group; Drug therapy group

SUMMARY:
This study is to examine whether the efficacy of DBT for BN is comparable with drug treatment, whether short-term and long-term efficacy of DBT combined with drug treatment of BN is better than single DBT or single drug treatment, and trying to explore predictable biological indicators of short-term and long-term efficacy of DBT for BN. Our study will use multi-center randomized controlled study design. 165 outpatients with BN will be recruited from Shanghai Mental Health Center, No.6 Hospital of Peking University and Shanghai Tongji Hospital. There will be three groups: DBT treatment group, Fluoxetine treatment group, DBT combined with fluoxetine treatment group. We prepare to recruit 165 patients with BN ,and each group is 55, and then three groups will be given standard intervention for 12 weeks. To assess the eating disorder symptoms, impulsive and emotional change, clinical symptom scales, psychological scales and the security indexs will be used at baseline, 4 weeks, 8 weeks, 12 weeks (end of treatment), 16weeks(1 month after treatment),24 weeks (3 months after treatment) and 36 weeks (6 months after treatment follow-up). Furthermore, brain MRI will be used for DBT treatment group at baseline, and 36 weeks.

DETAILED DESCRIPTION:
Bulimia nervosa(BN) is a chronic and refractory mental disorder characteristic of recurrent binge eating and weight control which mostly occur in adolescents and young women. The life-time prevalence ranges from 1.0%-4.2%, while in middle school and university, the prevalence can be 4.7-17%, and keep increasing. The recurrence rate of BN is also high, which can reach 25-63% six months after recovery. The nature cause can last several years showing a chronic feature. Patients with BN can also suffer from other severe psychosomatic complications, which harm the patients physical and mental health, thus lead to a mortality of 1% and negative impact on patients life and his/her family.

Antidepressant fluoxetine can reduce binge eating and purging behaviors in BN patients in a short time. It is the only drug approved by the US FDA for the treatment of BN, and also helps to prevent recurrence. However, there are still a considerable proportion of patients who keep a poor response to the medication. Cognitive behavioral therapy, Interpersonal therapy and other traditional psychotherapy are effective for BN patients, however, as many as 50% of BN patients still have ED symptoms. Therefore, it is necessary to develop a more effective new treatment method. Dialectical behavior therapy as a new and effective psychological therapy in the treatment of BN, proven to reduce binge eating, purging behaviors and non-suicidal act of self harm in adolescents and adults in foreign countries, now shows its superiority in the treatment of BN. At present, because of an acute shortage of psychotherapists in China, carrying out the DBT group is significant. However, currently there are no related research reports in china.

This study is to examine whether the efficacy of DBT for BN is comparable with drug treatment, whether short-term and long-term efficacy of DBT combined with drug treatment of BN is better than single DBT or single drug treatment, and trying to explore predictable biological indicators of short-term and long-term efficacy of DBT for BN. This study will use multi-center randomized controlled study design. 165 outpatients with BN will be recruited from Shanghai Mental Health Center, No.6 Hospital of Peking University and Shanghai Tongji Hospital. This study will use multi-center randomized controlled study design. 165 outpatients with BN will be recruited from Shanghai Mental Health Center, No.6 Hospital of Peking University and Shanghai Tongji Hospital. There will be three groups: DBT treatment group, Fluoxetine treatment group, DBT combined with fluoxetine treatment group. The investigator prepare to recruit 165 patients with BN ,and each group is 55, and then three groups will be given standard intervention for 12 weeks. To assess the eating disorder symptoms, impulsive and emotional change, clinical symptom scales, psychological scales and the security indexs will be used at baseline, 4 weeks, 8 weeks, 12 weeks (end of treatment), 16weeks(1 month after treatment),24 weeks (3 months after treatment) and 36 weeks (6 months after treatment follow-up). Furthermore, brain MRI will be used for DBT treatment group at baseline, and 36 weeks.

This study was designed with sufficient consideration about innovation as well as feasibility, and is to be operated on well proved theoretical basis and guidance of an operation manual. If successful, results of this study may bring great improvement to clinical practice of this refractory mental disorder.

ELIGIBILITY:
Inclusion Criteria:

* Female;
* Han nationality;
* Aged 18-40 years;
* right handedness;
* above primary education;
* met DSM-IV criteria for BN;

Exclusion Criteria:

* diagnosed with a mental illness;

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 101 (Actual)
Dates: Start 2018-06-13 (Actual); Primary Completion 2020-12-30 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
Eating Disorder Examination(EDE-Q) | Change from Baseline eating attitudes and behaviors at 4 weeks,8weeks,12weeks,36weeks,60weeks.
  EDE-Q can evaluate the eating disorder behavior and psychology characteristics and assess their frequency and intensity, which can assess the severity of eating disorders.

SECONDARY OUTCOMES:
Eating Disorder Inventory(EDI-II) | Change from Baseline eating attitudes, behaviors and pathologic psychological characteristics at 4 weeks,8weeks,12weeks,36weeks,60weeks.
  EDI-II can assess the eating attitudes and behaviors. It can evaluate the pathologic psychological characteristics of BN patients.
Barratt Impulsiveness Scale(BIS-II) | Change from Baseline the severity of impulse suppression orientation at 4 weeks,8weeks,12weeks,36weeks,60weeks.
  This tool can measure the severity of impulse suppression orientation.
Hamilton Depression Scale(HAMD) | Change from Baseline the severity of the symptoms of depression at 4 weeks,8weeks,12weeks,36weeks,60weeks.
  Measurement of the severity of the symptoms of depression.
Hamilton Anxiety Scale(HAMA) | Change from Baseline the severity of the symptoms of anxiety at 4 weeks,8weeks,12weeks,36weeks,60weeks.
  Measurement of the severity of the symptoms of anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: Jue Chen, PHD, Principal Investigator — Shanghai Mental Health Center
Locations (1):
- Shanghai Mental Health Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
The study protocol and baseline characteristics of participants
Supporting Information: Study Protocol, SAP
Time Frame: when we ended the experiment at 2019, we will share the data.
Access Criteria: DBT;Dialectical Behavioral Group Therapy; BN; Bulimia Nervosa

REFERENCES:
- [Background] Fischer S, Peterson C. Dialectical behavior therapy for adolescent binge eating, purging, suicidal behavior, and non-suicidal self-injury: a pilot study. Psychotherapy (Chic). 2015 Mar;52(1):78-92. doi: 10.1037/a0036065. Epub 2014 Apr 28. PMID 24773094
- [Background] Klein AS, Skinner JB, Hawley KM. Adapted group-based dialectical behaviour therapy for binge eating in a practicing clinic: clinical outcomes and attrition. Eur Eat Disord Rev. 2012 May;20(3):e148-53. doi: 10.1002/erv.2165. Epub 2012 Feb 24. PMID 22367862